CLINICAL TRIAL: NCT06449183
Title: Real-life Performance and Added Value of the VIDAS® TBI Blood Test in the Assessment of Mild Traumatic Brain Injury (mTBI), in Subjects with a Glasgow Coma Scale (GCS) Between 13-15
Brief Title: VIDAS® TBI Real Life Performance in Subjects with Mild Traumatic Brain Injury (mTBI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BM-2023-12
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-07

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Mild Traumatic Brain Injury; mTBI; TBI; Biomarkers; Automated assays; Ubiquitin Carboxy-terminal Hydrolase-L1 (UCH-L1); Glial Fibrillary Acidic Protein (GFAP); Canadian CT Head Rule; Canadian CT Head Rule (CCHR); Performance; Economic outcomes; Clinical outcomes; CT-Scan; Emergency Department (ED)
MeSH Terms: conditions — Brain Concussion; Emergencies

STUDY DESIGN:
Intervention Model Description: Single Prospective Cohort. Multicentric, International clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Subjects with Mild Traumatic Brain injury (Experimental): Subjects presenting to the ED within 12 hours of suspected mild head trauma and a Glasgow Score of 13-15 undergo to blood collection for VIDAS® TBI [GFAP, UCH-L1] testing.
  Interventions: Diagnostic Test: VIDAS® TBI Test [GFAP and UCH-L1 assays]

INTERVENTIONS:
Diagnostic Test: VIDAS® TBI Test [GFAP and UCH-L1 assays] — The VIDAS® TBI (GFAP, UCH-L1) test is composed of two automated assays - VIDAS® TBI (GFAP) and VIDAS® TBI (UCH-L1) - to be used on the VIDAS® family of instruments for the quantitative measurement of Glial 15 Fibrillary Acidic Protein (GFAP) and Ubiquitin C-terminal Hydrolase- L1 (UCH-L1) in human serum using the Enzyme Linked Fluorescent Assay (ELFA) technique. The results of both assays are required to obtain an overall qualitative test interpretation.

SUMMARY:
Decision Rules for an initial CT-scan in patients arriving to Emergency Department (ED) and presenting a mild traumatic brain injury could be optimized by the use of an objective parameter easily and rapidly measured. This may be the place for serum biomarkers providing a quick and accurate assessment. BioMérieux has now developed an automated assay for the measurement of serum Glial Fibrillary Acidic Protein (GFAP) and Ubiquitin C-terminal Hydrolase (UCH-L1), the VIDAS® TBI assay to fill out this unmet needs. The goal of the herein study is to generate real-world data and evidences to support the VIDAS® TBI performances.

DETAILED DESCRIPTION:
The assessment of severity of TBI patients is based on the Glasgow Coma Scale (GCS) and the initial management in the ED includes performing a non-contrast brain Computed Tomography (CT) scan if the patient meets specific conditions. To date, real world data show that EDs would actually not follow guideline recommendations and a substantial CT overuse is observed. Management strategies are becoming more and more focused on selective CT use to effectively manage health care resources. Efforts have been made to optimize the indications for brain CT scan after mTBI. Although brain CT scan plays a central role after mTBI, there is an unmet clinical need for an objective tool to optimize indications for CT scan, reduce patient radiation exposure, and possibly predict patient outcome. Clinical Decision Rules for an initial CT-scan could be optimized by the use of an objective parameter easily and rapidly measured. This may be the place for serum biomarkers providing a quick and accurate assessment. BioMérieux has now developed an automated assay for the measurement of serum Glial Fibrillary Acidic Protein (GFAP) and Ubiquitin C-terminal Hydrolase (UCH-L1), the VIDAS® TBI assay to fill out this unmet needs. The goal of the herein study is to generate real-world data and evidences to support the VIDAS® TBI performances.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject ≥ 18 years old
* Subject with a Glasgow Coma Scale (GCS) score between 13-15 on admission
* Subject presenting to the Emergency Department for suspected mild Traumatic Brain Injury
* Subject with a non-contrast head Computed Tomography (CT) scan ordered per the clinical site's care usual care
* Blood sampling possible within 12 hours of injury (1 tube of 4-5 mL of blood)
* Subject expected to stay at least 2 hours in the ED or in a ward
* Subject with signed Informed Consent Form (ICF)

Exclusion Criteria:

* Time of injury unknown
* Subject with non-traumatic neurological disorders (e.g, dementia, Parkinson's disease, multiple sclerosis, seizure disorder, brain tumors, spontaneous intracranial haematoma)
* Neurosurgery, stroke or transient ischemic attack within the last 30 days
* Subject with an active cancer
* Subject with penetrating head injury
* Special populations, including women with known pregnancy, prisoners, or institutionalized individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-06-16 (Estimated); Study Completion 2025-11-16 (Estimated)

PRIMARY OUTCOMES:
To determine VIDAS® TBI sensitivity to exclude the presence of an intracranial lesion | 12 hours post mild brain trauma
To determine VIDAS® TBI specificity to exclude the presence of an intracranial lesion | 12 hours post mild brain trauma
To determine VIDAS® TBI Positive Predictive Value to exclude the presence of an intracranial lesion | 12 hours post mild brain trauma
To determine VIDAS® TBI Negative Predictive Value to exclude the presence of an intracranial lesion | 12 hours post mild brain trauma
To determine VIDAS® TBI Positive Likelihood Ratio to exclude the presence of an intracranial lesion | 12 hours post mild brain trauma
To assess VIDAS® TBI Negative Likelihood Ratio to exclude the presence of an intracranial lesion | 12 hours post mild brain trauma

SECONDARY OUTCOMES:
To determine Canadian CT Head Rule specificity combined to VIDAS specificity to exclude the presence of an intracranial lesion | 12 hours post mild brain trauma
To determine Canadian CT Head Rule sensitivity combined to VIDAS sensitivity to exclude the presence of an intracranial lesion | 12 hours post mild brain trauma
To determine Canadian CT Head Rule Positive Predictive Value combined to VIDAS positive Predictive Value to exclude the presence of an intracranial lesion | 12 hours post mild brain trauma
To determine Canadian CT Head Rule Negative Predictive Value combined to VIDAS Negative Predictive Value to exclude the presence of an intracranial lesion | 12 hours post mild brain trauma
To determine Canadian CT Head Rule Negative Likelihood Ratio combined to VIDAS Negative Likelihood Ration to exclude the presence of an intracranial lesion | 12 hours post mild brain trauma
To determine Canadian CT Head Rule Positive Likelihood Ratio combined to VIDAS Positive Likelihood Ration to exclude the presence of an intracranial lesion | 12 hours post mild brain trauma
To estimate the impact of the use of VIDAS® TBI on the time to discharge | 3 months
To estimate the expected impact of the use of VIDAS® TBI on patient stay in the ED | 3 months
To estimate the expected impact of the use of VIDAS® TBI on hospitalization decision | 3 months
To estimate the expected impact of the use of VIDAS® TBI on time to medical decision | 3 months
To estimate the impact of the use of VIDAS® TBI on the patient's monitoring duration | 3 months
to measure the percentage of CT-scan potentially avoided | 3 months
To estimate the saving costs when using VIDAS® TBI in comparison with usual clinical sites' care. | 3 months
To estimate the costs of Length of stay in Emergency Department (ED) when using VIDAS® TBI in comparison with usual clinical sites' care. | 3 months
To estimate the associated costs of Length of stay in the hospital when using VIDAS® TBI in comparison with usual clinical sites' care. | 3 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Orlando Health, Orlando, Florida
  - Wayne State University, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of Rochester, Rochester, New York

IPD SHARING:
Plan to Share IPD: No